CLINICAL TRIAL: NCT00635232
Title: A Randomized, Double-Blind, Placebo And Active-Controlled, Parallel Group Study To Evaluate The Dose-Related Efficacy And Safety Of PS433540 In Subjects With Hypertension
Brief Title: A Study To Evaluate The Dose-Related Efficacy and Safety of PS433540 in Subjects With Hypertension
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PCO-C-006
Record Dates: First submitted 2008-03-06; First posted 2008-03-13 (Estimated); Results first posted 2011-09-13 (Estimated); Last update posted 2011-09-16 (Estimated); Status verified 2011-09

CONDITIONS: Hypertension
Keywords: Hypertension; High Blood Pressure
MeSH Terms: conditions — Hypertension | interventions — Irbesartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Irbesartan 300mg (Active Comparator): Irbesartan 300 mg once daily
  Interventions: Drug: irbesartan
- Placebo (Placebo Comparator): Blinded Placebo Treatment
  Interventions: Drug: placebo
- PS433540 200mg (Experimental): PS433540 200mg once daily
  Interventions: Drug: PS433540
- PS433540 400mg (Experimental): PS433540 400mg once daily
  Interventions: Drug: PS433540
- PS433540 800mg (Experimental): PS433540 800mg once daily
  Interventions: Drug: PS433540

INTERVENTIONS:
Drug: irbesartan — 300 mg (2 x 150 mg capsules) once daily for 12 weeks
  Other Names: Avapro
  Arms: Irbesartan 300mg
Drug: placebo — placebo capsules once daily for 12 weeks
  Arms: Placebo
Drug: PS433540 — 200 mg (2 x 100 mg capsules) once daily for 12 weeks
  Arms: PS433540 200mg
Drug: PS433540 — 400 mg (4 x 100 mg capsules) once daily for 12 weeks
  Arms: PS433540 400mg
Drug: PS433540 — 800 mg (8 x 100 mg capsules) once daily for 12 weeks
  Arms: PS433540 800mg

SUMMARY:
The purpose of this study is to learn which doses of PS433540 should be given to patients with high blood pressure to lower their blood pressure. This study will also examine how safe PS433540 is when taken by patients with high blood pressure. Approximately 720 patients will be evaluated so that about 375 patients will be entered into the treatment phase of the study and be given PS433540.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 18 - 70 years
* Mean seated Systolic Blood Pressure (SBP) ≥ 140 mmHg and < 180 mmHg and mean seated Diastolic Blood Pressure (DBP) > 90 and < 109 mmHg at two consecutive qualifying visits (Visits 3/3.5 and Visit 4). The mean difference in DBP between the two consecutive qualifying visits must be ≤ 10 mmHg.
* Women of child-bearing potential (WOCBP) must use two reliable forms of contraception if sexually active. Alternatively, female subjects must be postmenopausal (for at least 1 year).

Exclusion Criteria:

* Subjects with serious disorders which may limit the ability to evaluate the efficacy or safety of PS433540, including cardiovascular (includes subjects who are known to have coronary artery disease), renal (including the absence of one kidney), pulmonary, hepatic, gastrointestinal (including clinically significant malabsorption), endocrine/metabolic, hematologic, neurologic and psychiatric diseases.
* History of malignancy other than adequately treated basal cell or squamous cell skin cancer.
* Subjects with a history of myocardial infarction or New York Heart Association (NYHA) class II-IV heart failure.
* Subjects with a history of cerebrovascular accident or transient ischemic attack.
* Subjects with clinically significant cardiac conduction defects, including second or third degree Atrioventricular Block (AV block), left bundle branch block, sick sinus syndrome, atrial fibrillation, atrial flutter, an accessory bypass tract, or any arrhythmia requiring medication.
* Subjects with hemodynamically significant valvular disease.
* Subjects with history of type 1 diabetes mellitus and subjects with a history of type 2 diabetes mellitus using antihyperglycemic medication (oral medication, insulin, or exenatide) are excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rene Belder, MD, Study Director — Ligand Pharmaceuticals; Joel Neutel, MD, Principal Investigator — Orange County Research Center
Locations (40):
- United States (40):
  - Advanced Clinical Research 1000 Forrest Place Suite 2 Pell City, Pell City, Alabama
  - Premiere Pharmaceutical Research, LLC, Tempe, Arizona
  - Genova Clinical Research AZ, Tucson, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Associated Pharmaceutical Research Center, Buena Park, California
  - Clinical Trials Research CA, Lincoln, California
  - Long Beach Center for Clinical Research, Long Beach, California
  - National Research Institute, Los Angeles, California
  - Superior Regional Research, LLC, Sacramento, California
  - Orange County Research Center, Tustin, California
  - Westlake Medical Center, Westlake Village, California
  - Univ. Clinical Research Deland, LLC., DeLand, Florida
  - Allan Graff, Fort Lauderdale, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - North County Medical, Sebastian, Florida
  - Q Clinical Research, Decatur, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Cedar Crosse Research Center, Chicago, Illinois
  - Midwest Institute for Clinical Research, Indianapolis, Indiana
  - MD Medical Research, Oxon Hill, Maryland
  - Cary Medical Research, Cary, North Carolina
  - Metrolina Medical Research, Charlotte, North Carolina
  - Unifour Medical Research NC, Hickory, North Carolina
  - Northstate Clinical Research, Lenoir, North Carolina
  - Triangle Medical Research NC, Raleigh, North Carolina
  - Crescent Medical Research, Salisbury, North Carolina
  - New Hanover Medical Rersearch, Wilmington, North Carolina
  - Peidmont Medical Research Associates, Winston-Salem, North Carolina
  - The Lindner Center, Cincinnati, Ohio
  - Delaware Smith Clinic, Delaware, Ohio
  - Smith Clinic, Marion, Ohio
  - COR Clinical Research, L.L.C, Oklahoma City, Oklahoma
  - Brandywine Clinical Research Center, Downingtown, Pennsylvania
  - Hypertension & Nephrology Inc, Providence, Rhode Island
  - Punzi Medical Center, Carrollton, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - IMED Research PA, San Antonio, Texas
  - Hampton Roads Center for Clinical Research, Norfolk, Virginia
  - Gemini Scientific LLC, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All subjects were weaned off all antihypertensive medication prior to be entered into a 4-week single-blind placebo run-in period. Subjects had to have eligible Seated systolic and diastolic BP measurements during the single-blind placebo run-in phase to be eligible for the double blind portion of the study.
Period: Overall Study
Arm/Group | Irbesartan 300mg | Placebo | PS433540 200mg | PS433540 400mg | PS433540 800mg
Started | 58 | 59 | 58 | 58 | 28
Completed | 44 | 39 | 55 | 48 | 20
Not Completed | 14 | 20 | 3 | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Irbesartan 300mg | Placebo | PS433540 200mg | PS433540 400mg | PS433540 800mg | Total
Number analyzed (Participants) | 58 | 59 | 58 | 58 | 28 | 261
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 53 | 52 | 50 | 48 | 28 | 231
  >=65 years | 5 | 7 | 8 | 10 | 0 | 30
Age Continuous [Mean (Standard Deviation); unit: years] | 51.5 (8.97) | 54.2 (8.12) | 53.2 (10.58) | 53.4 (10.71) | 51.4 (9.92) | 52.9 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 27 | 26 | 17 | 123
  Male | 35 | 29 | 31 | 32 | 11 | 138
Region of Enrollment [Number; unit: participants]
  United States | 58 | 59 | 58 | 58 | 28 | 261

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Seated Systolic Blood Pressure (SBP) Following 12 Weeks of Treatment With PS433540 200 mg, 400 mg, 800 mg and Placebo.
Time Frame: 12 weeks
Population: The primary efficacy population was the Full Analysys Set (FAS) population= all randomized subjects who took at least one dose of the assigned study drug and had both baseline and post-baseline mean seated SBP. Both LOCF and observed-data set approach were performed.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Irbesartan 300mg | Placebo | PS433540 200mg | PS433540 400mg | PS433540 800mg
Number analyzed (Participants) | 58 | 59 | 58 | 58 | 28
mm Hg | -10.7 (14.32) | 1.8 (14.16) | -13.2 (13.61) | -14.2 (11.90) | -23.4 (18.70)

2. Secondary Outcome: Change From Baseline in Mean Seated Diastolic Blood Pressure (DBP) Following 12 Weeks of Treatment With PS433540 200 mg, 400 mg, 800 mg and Placebo.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Irbesartan 300mg | Placebo | PS433540 200mg | PS433540 400mg | PS433540 800mg
Number analyzed (Participants) | 58 | 59 | 58 | 58 | 28
mm Hg | -7.1 (9.19) | 0.2 (9.68) | -7.2 (8.34) | -9.2 (9.10) | -14.3 (10.53)

3. Secondary Outcome: The Percentage of Patients Treated With Each Dose of PS433540 Who Achieved Blood Pressure Control, Defined as <140/90 mmHg, After 12 Weeks of Treatment.
Time Frame: 12 weeks
Population: Full analysis set (LOCF)
Measure: Number; unit: participants
Arm/Group | Irbesartan 300mg | Placebo | PS433540 200mg | PS433540 400mg | PS433540 800mg
Number analyzed (Participants) | 58 | 59 | 58 | 58 | 28
participants | 17 | 5 | 21 | 28 | 16

ADVERSE EVENTS:
Arm/Group | Irbesartan 300mg | Placebo | PS433540 200mg | PS433540 400mg | PS433540 800mg
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/59 | 0/58 | 1/58 | 0/28
Other Adverse Events (participants affected / at risk) | 19/58 | 20/59 | 10/58 | 25/58 | 17/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Irbesartan 300mg (N=58) | Placebo (N=59) | PS433540 200mg (N=58) | PS433540 400mg (N=58) | PS433540 800mg (N=28)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — reported during the placebo run-in phase- subject not on active treatment at the time of report.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Irbesartan 300mg (N=58) | Placebo (N=59) | PS433540 200mg (N=58) | PS433540 400mg (N=58) | PS433540 800mg (N=28)
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 2
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 2
Dizziness (Nervous system disorders) | 2 | 2 | 0 | 2 | 3
Eye Disorders (Eye disorders) | 0 | 3 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 1 | 0 | 4 | 0
Feces Discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 0 | 1
Haemoglobin abnormal (Investigations) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 4 | 10 | 0 | 3 | 2
Hot Flush (Vascular disorders) | 0 | 0 | 0 | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1 | 2 | 1
Influenza (Infections and infestations) | 1 | 1 | 0 | 2 | 1
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 2 | 2 | 2 | 4 | 0
Migraine (Nervous system disorders) | 2 | 3 | 0 | 2 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 2
Oedema Peripheral (General disorders) | 2 | 1 | 2 | 4 | 3
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 2 | 1 | 2 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Tooth Abcess (Infections and infestations) | 1 | 0 | 0 | 2 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 2 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 3 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The 800mg dose level was discontinued from further enrollment per protocol amendment due to findings from another PS433540 trial that suggested clinical benefit beyond 500mg was expected to be limited.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No